CLINICAL TRIAL: NCT03791528
Title: Assessing the Effects of Kinesiological Taping On Function And Pain Scores in Patients With Sacroiliac Joint Dysfunction
Brief Title: Is Kinesio Taping Treatment Effective in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Assoc Prof, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DorkuzEUTuran
Record Dates: First submitted 2018-12-02; First posted 2019-01-02 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Sacroiliac Joint Dysfunction; Kinesio Taping Treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio-taping Treatment Group (Active Comparator): In treatment group; Kinesio-taping 3 times at 5-day intervals, one of the fan-shaped cut bands, 2-3 inches above the sacroiliac joint (SIJ), and the other below 2-3 inches below the SIJ, and crossed each other by 90 degrees. evaluated at baseline, the twentieth minute after application and on the 15th day by physical examination of the sacroiliac joint, visual analog scale, Modified Oswestry Low Back Pain Disability Questionnaire
  Interventions: Other: Kinesio-taping treatment group
- Control Group (No Intervention): Without Kinesio-taping treatment evaluated at baseline and on the 15th day by physical examination of the sacroiliac joint, visual analog scale, Modified Oswestry Low Back Pain Disability Questionnaire

INTERVENTIONS:
Other: Kinesio-taping treatment group — In treatment group; Kinesio-taping 3 times at 5-day intervals, one of the fan-shaped cut bands, 2-3 inches above the SIJ, and the other below 2-3 inches below the SIJ, and crossed each other by 90 degrees. evaluated at baseline, the twentieth minute after application and on the 15th day by physical examination of the sacroiliac joint, visual analog scale, Modified Oswestry Low Back Pain Disability Questionnaire.
  Arms: Kinesio-taping Treatment Group

SUMMARY:
Low back pain is a common condition that affects 70% of people at least once. Sacroiliac joint Dysfunction (SIJD) is a skipped health problem that is ignored in patients with low back or hip pain. Fluoroscopy-guided SIJ injection showed that SIJD is a source of pain in 13-30% of patients with chronic low back pain. Inadequate function of SIJ leads to abnormal gait pattern, pain during walking, increase in load on discs, long-term interdisciplinary stability and causing to increase of the listhesis. The pain worsens with running, climbing stairs or standing up from the sitting position. Pharmacological, non-pharmacological and if required surgical treatment may be applied in the osteoarthritis treatment. Non-pharmacological treatment includes patient education, exercise, massaging, SIJ, manipulation-mobilization, chiropractic applications, physical therapy modalities, use of the assistive device.

Kinesio Taping is a treatment that has not been studied much and can be applied in SIJD. When investigators reviewed the literature, investigators found a study and a case report investigating the activity of Kinesio taping in sacroiliac joint dysfunction. Although the mechanism of Kinesio taping cannot be understood, it is claimed that it has four beneficial effects: normalizes muscular function, improves blood and lymphatic circulation, reduces pain, regulates possible disorders of joints. In studies showing the effectiveness of Kinesio banding in the reduction of pain in health problems related to the waist area with the highest number of publications, it was noted that the pain was reduced rapidly within three days, decreased the need for analgesics within two weeks and increased function in daily living activities.

DETAILED DESCRIPTION:
The study is a randomized, controlled study. 52 participants will be included to study who apply to Dokuz Eylül University Faculty of Medicine, Department of Physical Medicine and Rehabilitation Clinic with the complaint of hip and back pain, aged between 18-60 years. Participants have diagnosed as Sacroiliac Joint Dysfunction according to The International Association for the Study of Pain (IASP) diagnostic criteria. These participants will be divided into two groups randomly (Treatment group n:26, control group n:26). Because the therapeutic effect may be seen with unsealed banding in Kinesio taping and the placebo effect may not be evaluated, After the last evaluation, participants in both groups will be given the necessary treatment and since there is no study on this subject in the literature, no treatment was given to the control group due to the fact that the actual effect of banding was desired. The treated group received Kinesio taping 3 times at 5-day intervals, one of the fan-shaped cut bands, 2-3 inches above the SIJ, and the other below 2-3 inches below the SIJ, and crossed each other by 90 degrees. Both groups were evaluated at baseline and on the 15th day by physical examination of the sacroiliac joint, visual analog scale, Modified Oswestry Pain Inquiry Form. The kinesiological taping group was also evaluated with VAS and positive SIJ pain provocation tests, 20 minutes after the first banding, to assess the acute effect.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-60
2. Based on the diagnostic criteria proposed by the International Association for the Study of Pain (IASP):

   i.Pain in the SIE region (hip/groin or lower extremity) ii.The pain felt in SIS, revitalized by specific provocation tests
3. Patients with sacroiliac joint dysfunction and validity-validity-tested provocation tests, at least 3 of 6 tests are positive

1.Distraction 2.Compression 3.Gaenslen 4.POSH Test ( Thigh Thrust) 5.Sacral Push 6.FABER 4. Patients excluded from the presence of sacroiliitis by previous examinations and examinations 5. The signing of the informed consent form

Exclusion Criteria:

1. Severe cognitive dysfunction
2. The presence of a neurological deficit in the lower extremity
3. Presence of known central nervous system or peripheral nervous system disease
4. Presence of known rheumatic disease (rheumatoid arthritis, ankylosing spondylitis, etc.)
5. Have undergone major surgery for lower back and waist
6. Pregnancy
7. Spondylolisthesis
8. Built-in osteoporosis
9. The presence of malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS ) for sacroiliac pain | Change from baseline pain score at 15 th day
  visual analog scale, 0 minimum, 10 maximum score, higher values represent a worse outcome.

SECONDARY OUTCOMES:
Modified Oswestry Pain Inquiry Form for pain and quality of life | All patients will evaluated at baseline, twentieth minute after application and on the 15th day.
  It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Dilek, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided